CLINICAL TRIAL: NCT07297511
Title: The Application of Vertical Jump Performance in Return-to-Play Assessment for Anterior Cruciate Ligament Reconstruction Athletes
Brief Title: Application of Multiple Vertical Jump Tests in Return-to-Play Assessment for Anterior Cruciate Ligament Reconstruction Athletes
Acronym: RTP-VJ
Status: Not yet recruiting | Type: Observational
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Cheng-Yen Teng, Principal Investigator, Kaohsiung Medical University
Other Study IDs: KMUHIRB-F(II)-202 20046; KMUHIRB-F(II)-202 20046 (Other: Kaohsiung Medical University Chung-Ho Memorial Hospital Institutional Review Board)
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-07

CONDITIONS: ACL Reconstruction
Keywords: ACL reconstruction; vertical jump test; return to play

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health: Control group: The group include athletes with no lower limbs injury.Participants must be aged 18-35 years and must be elite athletes who have competed in national-level competitions.
- ACL reconstruction: Participants must be aged 18-35 years with unilateral ACL rupture confirmed by MRI, Lachman test grade ≥2, and reconstruction using hamstring or gracilis autograft with at least 6 months post-operative. Participants must have completed rehabilitation with clearance from an orthopedic surgeon or physical therapist, demonstrate no other lower extremity injuries, and have no contralateral lower limb injury within the past 3 months. Additionally, quadriceps strength symmetry index must be ≥90%, and participants must be elite athletes who have competed in national-level competitions.

SUMMARY:
Anterior cruciate ligament (ACL) injury is a common sports-related injury, particularly in sports that require extensive jumping and cutting movements. Although anterior cruciate ligament reconstruction (ACLR) surgery can restore knee stability, many athletes still face the risk of re-injury after returning to competition.Current return-to-play assessment relies primarily on single-plane horizontal hop tests and symmetry indices (LSI ≥ 90%); however, an increasing body of research suggests that these tests may not comprehensively reflect functional deficits in the vertical plane, repeated hopping, or high-intensity sport-specific activities.This study hypothesizes that incorporating multiple vertical jump tests-including single-leg vertical jumps and 10-second repeated vertical jumps-combined with advanced force plate analytics (such as Reactive Strength Index [RSI] and Time to Stabilization [TTS])-can more sensitively reveal residual neuromuscular control deficits following surgery. This approach would provide evidence-based guidance for return-to-play decision-making, thereby improving athletes' long-term athletic performance and safety.

DETAILED DESCRIPTION:
This cross-sectional study compares biomechanical performance between ACLR athletes (>6 months post-op) and healthy controls to evaluate whether vertical jump protocols reveal greater limb asymmetries compared to traditional horizontal hop tests. Following a 5-minute stationary bicycle warm-up and familiarization trials, participants perform four unilateral tasks on both limbs: Single-Legged Hop for Distance (SHD), Crossover Hop for Distance (CHD), Single-Legged Vertical Countermovement Jump (SLVJ), and 10-Second Repeated Single-Legged Vertical Jump (SLVJs). All tasks are performed with hands on hips to minimize compensatory motion. Three successful trials are recorded per limb per task with 3-minute rest intervals between sets. Trials are discarded if participants land on the contralateral limb, lose balance, or fail to land on the force plate. Vertical ground reaction forces are collected using a dual-force plate system (Hawkin Dynamics, 3rd Generation) at 1000 Hz. Data processing calculates Limb Symmetry Index (LSI), Modified Reactive Strength Index (RSI) from SLVJs as Jump Height divided by Movement Time, Time to Stabilization (TTS) defined as the duration for vGRF to stabilize within ±5% of body weight, and eccentric/concentric impulse.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age 18-35 years

  2.Unilateral anterior cruciate ligament (ACL) rupture confirmed by magnetic resonance imaging (MRI)

  3.Positive Lachman test grade ≥2 pre-operatively

  4.Anterior cruciate ligament reconstruction (ACLR) using hamstring or gracilis autograft

  5.Post-operative time ≥6 months

  6.Completed rehabilitation program with clearance from orthopedic surgeon or physical therapist

  7.Quadriceps strength symmetry index ≥90%

  .Elite athlete status (prior participation in national-level competitions)

Exclusion Criteria:

1. Other lower extremity injuries or pathologies (including other knee ligament injuries)
2. Contralateral lower limb injury within the past 3 months
3. Quadriceps strength symmetry index <90%
4. Non-elite athlete status (no prior national-level competition participation)
5. Incomplete rehabilitation or lack of medical clearance

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of two distinct groups: (1) ACLR athletes: elite athletes aged 18-35 years who have undergone unilateral anterior cruciate ligament reconstruction using hamstring or gracilis autograft with a minimum of 6 months post-operative. These participants will be recruited from orthopedic clinics, sports medicine centers, and rehabilitation facilities in the region. (2) Healthy controls: age, sex, and athletic-level matched individuals aged 18-35 years with no history of lower extremity injuries, recruited from local athletic facilities, university sports programs, and community sports organizations. Both groups must have elite athlete status, defined as prior participation in national-level sports competitions. The ACLR group represents athletes in the late rehabilitation phase preparing for return-to-play, while the healthy control group serves as a reference for normal biomechanical performance.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Limb asymmetry index,LSI | At baseline (single testing session; no longitudinal follow-up)
  Limb Symmetry Index (LSI) calculated as (|Uninvolved limb value - Involved limb value| / (Uninvolved limb value + Involved limb value)) × 100% for each of the four jump tasks: Single-Legged Hop for Distance (SHD), Crossover Hop for Distance (CHD), Single-Legged Vertical Countermovement Jump (SLVJ), and 10-Second Repeated Single-Legged Vertical Jump (SLVJs). LSI values will be compared between ACLR athletes and healthy controls to determine whether vertical jump protocols reveal greater limb asymmetries than traditional horizontal hop tests. Primary analysis will examine whether LSI differences in vertical jump tasks are statistically significantly lower (indicating greater asymmetry) than horizontal hop tasks, revealing residual neuromuscular deficits not detected by conventional return-to-play assessment.

SECONDARY OUTCOMES:
Modified Reactive Strength Index | At baseline (single testing session; no longitudinal follow-up)
  Modified Reactive Strength Index (mRSI) calculated as Flight Time(s) divided by Time to Take-off(s) for the 10-Second Repeated Single-Legged Vertical Jump (SLVJs) task.
Time to Stabilization (seconds) | At baseline (single testing session; no longitudinal follow-up)
  Time to Stabilization (TTS) measured during the Single-Legged Vertical Countermovement Jump (SLVJ) task, defined as the time required for vertical ground reaction force (vGRF) to return to and stabilize within ±5% of the participant's body weight following landing.
Single-Legged Hop for Distance (centimeter) | At baseline (single testing session; no longitudinal follow-up)
  Single-Legged Hop for Distance (SHD) measured as the maximum horizontal distance(centimeter) achieved during a single maximal hop on the tested leg, performed bilaterally.
Crossover Hop for Distance (centimeter) | At baseline (single testing session; no longitudinal follow-up)
  Crossover Hop for Distance (CHD) measured as the total horizontal distance covered during three consecutive hops crossing a centerline, performed bilaterally with emphasis on stability and continuity.
Jump Height(meter) | At baseline (single testing session; no longitudinal follow-up)
  Jump Height measured during the Single-Legged Vertical Countermovement Jump (SLVJ) and 10-Second Repeated Single-Legged Vertical Jump (SLVJs) tasks, calculated from the flight time (time from takeoff to landing) using force plate data.

CONTACTS AND LOCATIONS:
Overall Officials: GUO L Y Professor and Dean of college, Ph.D., Study Chair — Department of Sports Science, Kaohsiung Medical University, Taiwan
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the main published results, including demographic characteristics and biomechanical outcome measures (e.g., jump height, limb symmetry index, RSI, TTS, and impulse), will be shared with qualified researchers upon reasonable request, after approval of a data use agreement and in accordance with applicable ethical and regulatory requirements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified individual participate data (IPD) and supporting information will be available starting 2 years after the publication of the primary study results and will remain accessible for 5 years.
Access Criteria: The related supporting documents will only be made available to qualified researchers affiliated with academic institutions, medical organizations, or public health agencies. Applicants must submit a detailed research proposal and ethical approval documents, and access will be granted only upon approval.